CLINICAL TRIAL: NCT03381989
Title: Bioprosthetic or Native Aortic Scallop Intentional Laceration to Prevent Latrogenic Coronary Artery Obstruction (BASILICA)
Brief Title: Bioprosthetic or Native Aortic Scallop Intentional Laceration to Prevent Iatrogenic Coronary Artery Obstruction (BASILICA) Prospective Investigation
Acronym: BASILICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 999918018; 18-H-N018
Record Dates: First submitted 2017-12-21; First posted 2017-12-22 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-09

CONDITIONS: Native and Valve in Valve Aortic Valve Failure
Keywords: TAVR; Native Aortic Valve Failure; Valve in Valve Aortic Valve Failure; TAVR Associated Coronary Artery Obstruction; Electrosurgery
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single arm: open-label treatment (Experimental): The BASILICA procedure has three steps: (1) leaflet traversal with a guidewire, followed by (2) leaflet laceration, immediately followed by (3) TAVR.
  Interventions: Device: ASHI_INTECC Astato XS 20 0.014 guidewire

INTERVENTIONS:
Device: ASHI_INTECC Astato XS 20 0.014 guidewire — A coaxial traversal guiding catheter system (typically tandem catheters) directs electrosurgery devices (typically a rigid 0.014 guidewire inside a polymer jacket wire convertor) against the base of the coronary cusp targeted for laceration, using fluoroscopic and/or echocardiographic guidance. Traversal is accomplished by transcatheter electrosurgery by connecting the back end of the 0.014 guidewire to an electrosurgery pencil during short bursts of pure, cutting radiofrequency energy at ap-proximately 30W. The guidewire is repositioned as needed until it crosses the aortic leaflet and is snare-retrieved and externalized. Laceration is performed by positioning the laceration surface along the intended leaflet base, and applying tension on both free ends of the guidewire while simultaneously apply electrosurgery energy (typically 70W) in short bursts, until the laceration is complete and the guidewire is free.

SUMMARY:
Background:

TAVR is a common therapy for people with heart problems. It stands for transcatheter aortic valve replacement, TAVR can be a better option than surgery. But it isn t safe for everyone. It may block the arteries that supply blood to the heart muscle by pushing heart valve tissue outward. Researchers want to study a method that may make TAVR safer. It is known as Bioprosthetic or native Aortic Scallop Intentional Laceration to prevent Iatrogenic Coronary Artery obstruction (BASILICA).

Objective:

To study the feasibility and safety of BASILICA in people at high risk of coronary artery obstruction that complicates TAVR.

Eligibility:

People at least 21 years old whose heart doctors do not think they can have TAVR safely

Design:

Participants will be screened by a team of heart specialists. They will have heart and blood tests. They will answer questions.

Participants will have TAVR using BASILICA.

They will get general anesthesia or they will be sedated.

While using x-rays and echocardiography, doctors will cross and split the aortic valve leaflet using an electrified wire.

A standard TAVR valve will be implanted.

After the procedure, participants will have blood tests and physical exams. They will answer questions. They will have heart tests.

Participants will have a scan within 1 month and after 12 months. They will have heart tests during follow-up visits in the first year.

Sponsoring Institute: National Heart, Lung and Blood Institute

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) is an option to treat aortic valve stenosis or failure of a surgically implanted tissue valve. Sometimes TAVR displaces the diseased aortic valve leaflets outwards, causing life-threatening obstruction of the coronary arteries that supply blood to the heart. This is more common in surgically implanted tissue valves that are designed to achieve the largest aortic valve orifice area. Despite attempts to protect the coronary arteries from obstruction in these patients using coronary stents, the mortality of TAVR-associated coronary artery obstruction remains prohibitively high.

The investigators have developed and tested a technique to tear the existing aortic valve leaflet and enable TAVR in such patients. The procedure is called Bioprosthetic or native Aortic Scallop Intentional Laceration to prevent Iatrogenic Coronary Artery obstruction (BASILICA).

The purpose of this study is to perform BASILICA in patients who have no good options to prevent coronary artery obstruction during TAVR.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults age greater than or equal to 21 years
* High or extreme risk of surgical aortic valve replacement according to the local multidisciplinary heart team
* Undergoing TAVR for valve-in-valve or native aortic valve failure ( on-label TAVR)
* Deemed likely to suffer coronary artery obstruction from TAVR according to multidisciplinary heart team
* Concurrence of the study eligibility committee

EXCLUSION CRITERIA:

* Subjects unable to consent to participate, unless the subject has a legally authorized representative
* Excessive target aortic leaflet calcification or masses on baseline CT
* Survival despite successful procedure expected < 12 months
* Planned concurrent valve intervention in the same setting (such as transcatheter mitral valve therapy or paravalvular leak therapy)
* Subjects unwilling to participate or unwilling to return for study follow-up activities.
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (4):
- United States (4):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Khan JM, Greenbaum AB, Babaliaros VC, Dvir D, Reisman M, McCabe JM, Satler L, Waksman R, Eng MH, Paone G, Chen MY, Bruce CG, Stine AM, Tian X, Rogers T, Lederman RJ. BASILICA Trial: One-Year Outcomes of Transcatheter Electrosurgical Leaflet Laceration to Prevent TAVR Coronary Obstruction. Circ Cardiovasc Interv. 2021 May;14(5):e010238. doi: 10.1161/CIRCINTERVENTIONS.120.010238. Epub 2021 May 18. PMID 34003670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 participants enrolled on protocol. 30 started the protocol, after 1 participant withdrew consent prior to the procedure.
Period: Overall Study
Arm/Group | Single Arm: Open-label Treatment
Started | 30
Completed | 22
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm: Open-label Treatment
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure Success, Measured at Exit From the Catheterization Laboratory
Description: Successful BASILICA traversal and laceration; immediate survival; successful first TAVR device implantation; absence of coronary artery obstruction; and freedom from emergency cardiac surgery or reintervention related to the BASILICA or TAVR procedure.
Time Frame: 1 day
Population: Subjects who underwent the BASILICA procedure
Measure: Number; unit: participants
Arm/Group | Single Arm: Open-label Treatment
Number analyzed (Participants) | 30
participants | 28

2. Primary Outcome: Number of Participants Were Safety Endpoint is Freedom From Major Adverse Clinical Events (MACE)
Description: Freedom from major adverse clinical events (MACE) according to Valve Academic Research Consortium (VARC-2) at 30days.
Time Frame: 30 days
Population: Subjects who underwent the BASILICA procedure
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: Open-label Treatment: The BASILICA procedure has three steps: (1) leaflet traversal with a guidewire, followed by (2) leaflet laceration, immediately followed by (3) TAVR.Laceration of the aortic valve leaflet using electrosurgery energy.
Arm/Group | Single Arm: Open-label Treatment
Number analyzed (Participants) | 30
Participants | 21

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Single Arm: Open-label Treatment
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: Open-label Treatment (N=30)
Cardiac pacemaker insertion (Cardiac disorders) | 2
Hemodynamic instability from lacertation requiring vasopressors (Cardiac disorders) | 2
Secondary myocardial infarction (Cardiac disorders) | 1
Life threatening bleeding (Injury, poisoning and procedural complications) | 2 — not related to BASILICA
Major vascular complication (Injury, poisoning and procedural complications) | 6 — not related to BASILICA
Ischemic stroke (Nervous system disorders) | 3 — Disabling 1 subject Non-disabling 2 subjects
AKI - Acute Kidney Injury Stage 2/3 (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT03381989/Prot_SAP_000.pdf